CLINICAL TRIAL: NCT05096624
Title: Impact of Complete Removable Prosthetic Rehabilitations Performed by an Innovative DDTENS Protocol, on the Quality of Masticatory Function and the Management of Completely Edentulous Patients
Acronym: DD-TENS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RECHMPL20_0407
Record Dates: First submitted 2021-10-15; First posted 2021-10-27 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Disorder of Maxillary and Mandibular Dental Arch Relationship
Keywords: Total bimaxillary edentulous patient; Digital Denture; Neuromuscular occlusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DD-TENS (Digital Denture-Transcutaneous Electrical Nerve Stimulation) (Experimental): Patient with Complete Removable Prostheses according to DD-TENS system
  Interventions: Other: DD-TENS system
- Gold standard (Active Comparator): Patient with Complete Removable Prostheses according to usual care
  Interventions: Other: Gold Standard
- Digital denture System (Active Comparator): Patient with Complete Removable Prostheses according to Digital Denture system
  Interventions: Other: Digital Denture system

INTERVENTIONS:
Other: DD-TENS system — Use of DD-TENS system
  Arms: DD-TENS (Digital Denture-Transcutaneous Electrical Nerve Stimulation)
Other: Gold Standard — Gold standard
  Arms: Gold standard
Other: Digital Denture system — Use of Digital Denture system
  Arms: Digital denture System

SUMMARY:
Total edentulism is a profound physical, psychic and social handicap, which affects 5 million people in France. The most frequent complaint of edentulous patients rehabilitated by conventional Complete Removable Prostheses (CRP) is the reduction of masticatory efficiency. This alteration has medical repercussions and a negative psychological and social impact.

Our study aims to evaluate the impact of an innovative protocol on the quality of masticatory function, prosthetic treatment and, in fact, on the quality of life of the totally edentulous patient. This protocol combines the Digital Denture system with the transcutaneous electrical neurostimulation system (TENS®), in order to improve the balance of the dento-dental contacts of CRP. This new protocol is called DDTENS.

The first objective of the study is to compare the activity and balance of the masticatory muscles at 1 month (T1) of wearing the prostheses, between an experimental group benefiting from a CRP by the DDTENS protocol and 2 reference groups ( the first benefiting from a CRP by the conventional procedure and the second by the Digital Denture procedure) in bimaxillary total edentulous patients

The secondary objectives are:

* to compare the number of sessions required to obtain a finalized bimaxillary total removable prosthesis between the 3 groups.
* to compare the quality of life of patients with their CRP between the 3 groups, at 1 month and 4 months of wearing the prostheses.
* to compare the activity and balance of the masticatory muscles when the prostheses were put in the mouth (T0) and at 4 months (T4) of wearing the prostheses

The study design is a randomised open-label controlled pilot study with blinded reviewer assessment comparing 3 parallel groups:

* Experimental group: 10 bimaxillary edentulous patients rehabilitated by CRP using the DDTENS protocol.
* Control group 1: 10 edentulous bimaxillary patients rehabilitated by CRP according to the conventional method (gold standard technique).
* Control group 2: 10 edentulous bimaxillary patients rehabilitated by CRP using the Digital Denture procedure.

The expected benefits for patients in the DDTENS experimental group are the optimization of occlusal balance, the optimization of the time of integration of the prosthesis in the mouth, the time saving in the prosthetic treatment of the edentulous patient and the improvement of eating behaviours and quality of life of edentulous patients which would delay the entry of our patients into the sphere of dependence.

These results would allow the validation of a new rehabilitation protocol for the edentulous patient, leading to a modification of clinical practices.

DETAILED DESCRIPTION:
EPIDEMIOLOGY Total edentulism is defined by the total absence of teeth. It can be uni or bimaxillary and represents a profound physical, psychic and social handicap, affecting 5 million people in France. Despite progress in prophylaxis, the number of patients with total edentulism is constantly increasing.

There are several explanations for this phenomenon in France:

* Increase in life expectancy According to INSEE, life expectancy in France will increase from 75.2 years to 89.5 years for men and from 82.7 to 93 years for women between 2000 and 2050.
* Social precarity Social precarity is a societal problem that explains the delay or lack of dental care, leading to a higher rate of total edentulism among the most disadvantaged social class populations. Lifestyle behaviors such as smoking and alcohol consumption worsen this situation.
* Ageing of the population The arrival of the baby boomers in the 60+ age group and the increase in life expectancy explain the inevitable ageing of the population (3). People aged over 60 are expected to represent 1/3 of the population in 2050, whereas in 2005 they represented only 1/5.

This ageing is often associated with an alteration in physical and intellectual faculties. The relative well-being of 60-75 year old is gradually giving way to frailty. The challenge is to care for increasingly elderly edentulous patients. It is therefore essential to develop prosthetic rehabilitation practices to improve patient comfort.

Adopting an adapted treatment by limiting the number of appointments while maintaining an optimal quality of care is one of the objectives of our project.

PROBLEMATIC OF TOTAL EDENTULISM In the totally edentulous patient, certain physiological functions are altered (mastication, swallowing, taste, phonation). The most frequent complaint of edentulous patients rehabilitated by conventional Complete Removable Prosthesis (CRP) is the decrease in masticatory capacity. The masticatory capacity of edentulous patients is equivalent to 1/6 of dentate patients, not to mention the changes in eating behavior with certain foods banned from daily life.

This observation has medical repercussions (nutritional deficiencies, change in eating behavior, risk of misdirection, etc.) and a harmful psychological and social impact.

STATUS OF THE ISSUE Chewing ability can be understood by the shape of the chewing cycle, by bite force or by chewing efficiency. Studies have confirmed that conventional CRP do not restore optimal and efficient masticatory function, due to a lack of precision in the fabrication of the prosthesis and the empirical phase of occlusal balancing. Indeed, the dento-dental contacts, governed by the prosthetic mounting of the teeth, have a major impact on the functioning of the manducatory system.

These functional deficiencies can lead to a loss of physical and psychological autonomy, the gateway to iatrogenic dependence of the elderly in our hospitals.

How to improve masticatory efficiency in the totally edentulous patient? The placement of implants can be an alternative to remedy the problem of CRP retention, but the implant solution is not always feasible.

How to improve masticatory efficiency in the totally edentulous patient without the help of implants? The prosthetic equilibrium of an osteo-muco-portal prosthesis without implants is intimately linked to the tissue equilibrium and the neuro-musculo-articular equilibrium. Conversely, an unstable prosthesis leads to tissue damage and joint disorders.

The stability of the prosthesis is linked to the occlusal balance, the balance of the dento-dental contacts between the two arches. The complexity of the treatment lies in the determination of the inter-arch relationship or maxillo-mandibular relationship (MMR), in the vertical and horizontal directions. Indeed, in the totally edentulous patient, we have no reference points. The only usable determinants are the temporomandibular joints (TMJ).

To date, the conventional therapy or gold standard technique used for the rehabilitation of the totally edentulous patient, consists in recreating a "prosthetic substitution normality" by recording the maxillo-mandibular relationship, by putting the mandible in a reproducible position: the position of centered relation. The definition of the National College of Occlusodontics in 2001 tells us that it corresponds "to the condylar reference situation corresponding to a high, simultaneous condylo-disco-temporal coaptation obtained by non forced control. It is reproducible in a given time and for a given body posture and recordable from a mandibular rotation movement". The problem is that the TMJ is rarely healthy resulting in a more or less empirical and operator-dependent mandibular position. Errors in recording the mandibular position result in a loss of accuracy and an increased number of adjustment sessions.

In 2020, the use of digital tools aims to optimize and improve the recording of useful clinical data, the design and manufacture of a sustainable CRP. At present, no consensus exists but 2 paradigms coexist: the partial use of the digital tool, which punctuates the conventional steps and the use of protocols built entirely around the digital tool. These protocols have emerged secondarily and propose complete systems in 2 or 4 sessions.

Computer Aided Design and Manufacturing (CADCAM) systems applied to the rehabilitation of the totally edentulous patient are called Digital Denture protocols. Although CAD/CAM is a digital tool that has been used for many years in dentistry for the dentate patient, the Digital Denture system is not very widespread at the moment. This system ensures a better adaptation of the complete removable prostheses, thanks to the type of manufacture of the prostheses by machining, and a saving of time during the realization of the prostheses.

All in all, there is still the problem of the precision of the recording of the maxillo-mandibular relationship, which can lead to a number of additional adjustment sessions.

From these clinical findings, the two issues of this project were born:

1. How to improve the registration of the maxillomandibular relationship and the accuracy of occlusal balance?
2. How to reduce the number of adjustment sessions? Ultimately, the answer to these problems would influence the quality of the masticatory function and consequently the quality of life of the totally edentulous person.

INNOVATION The idea of the DDTENS protocol came from the reflection on the dentate patient with cranio-mandibular dysfunctions. Indeed, a transcutaneous electrical neurostimulation system (TENS®) is used in this clinical case, which allows muscular relaxation and the optimization of dento-dental contacts and thus the rebalancing of bilateral muscular forces.

The innovation consists in setting up an innovative protocol combining 2 existing systems: the Digital Denture system and a neuromuscular and electromyographic approach, via the transcutaneous electrical neurostimulation system (TENS®), in order to improve the registration and balance of dento-dental contacts in CRP.

HYPOTHESIS

1. Non-operator depending on the maxillo-mandibular relationship recording with a neuro-musculo-articular reference.
2. Reduction in the number of sessions for adjusting the prosthesis.
3. Optimization of the prosthetic treatment of edentulous patients.
4. Improvement of the occlusal balance and therefore of the quality of the masticatory function of edentulous patients (improvement of mastication, of eating behaviors (impact on nutrition, digestion, etc.), making it possible to delay the entry of our patients into the sphere of dependence.

OBJECTIVES

* Compare, within the framework of a randomized controlled pilot study, the activity and balance of the masticatory muscles at 1 month (T1) of wearing the prostheses, measured by a digital system combining electronic recording of mandibular movements and surface electromyography (K7 Evaluation System®), between an experimental group benefiting from a CRP by the DDTENS protocol and 2 reference groups: the first group benefiting from the performance of a CRP by the conventional procedure and the second by the Digital Denture procedure, in bimaxillary total edentulous patients
* Compare between the 3 groups, the number of sessions necessary to obtain a finalized prosthesis (prostheses are considered finalized when the prostheses worn by the patient are occlusally balanced and do not cause any mucosal injury).
* Compare the quality of life of patients with their PRC (assessment of chewing power, eating behavior, etc.), between the 3 groups, at 1 month and 4 months of wearing the prostheses.
* Compare, between the 3 groups, the activity and balance of the masticatory muscles when the prostheses are put in the mouth (T0) and at 4 months (T4) of wearing the prostheses.

METHODOLOGY The study design is a randomised, open-label, controlled pilot study with blinded reviewer evaluation comparing 3 parallel groups (2 control group and 1 experimental group).

The number of subjects to be included is 30. The randomization will be centralized (Ennov clinical software) and stratified by minimization on sex and age (60-69 and 70-85 years).

The masticatory muscle activity and balance are measured by a digital system combining electronic recording of mandibular movements and surface electromyography system (K7 Evaluation System®)

* Measurement of muscle activity = measurements will be made for all muscles at rest with and without prostheses.
* Muscle balance analysis = comparison of right and left muscle activity.
* Analysis of the chronology of muscle contraction on the right and left = muscle contraction symmetry

The number of sessions required to obtain a finished prosthesis recorded for each patient is listed.

The quality of life of the patients is assessed using a specific oral health measurement questionnaire (GOHAI). The GOHAI includes 12 items with 3 sub-dimensions (functional, psycho-social and pain/discomfort).

For each assessment (inclusion visit, 1-month post completion visit and 4-month post completion visit), the 3 sub-dimensions will be analyzed.

The patient must answer the 12 questions with "Never", "Rarely", "Sometimes", "Often" or "Always" (only one answer possible). Each answer is scored from 5 to 1 in this order, except for questions 3, 5 and 7 where the values are reversed. The associated total score varies from 12 to 60. The higher the score, the better the oral quality of life. The score obtained is classified into three categories:

12< <50: poor oral quality of life 51< <56: average oral quality of life 57< <60: good oral quality of life

ANTICIPATED BENEFITS AND RISKS

The expected benefits for patients in the TENS experimental group are:

* Optimization of maxillomandibular relationship registration
* Optimization of occlusal balance and masticatory functions (dental and muscular)
* Optimization of the integration time of prostheses in the mouth
* Improvement of the eating behaviors and quality of life of edentulous patients
* Time saving in the prosthetic treatment of the edentulous patient

The expected risks are:

* Muscle fatigue during TENS sessions if the application time is longer than 60 minutes.
* Number of adjustment sessions equivalent to the current Digital Denture protocol.

EXPECTED RESULTS AND PERSPECTIVES These results would allow the validation of a new gold standard protocol for the rehabilitation of the edentulous patient, leading to a modification of clinical practices.

Perspectives : This study could serve as the basis for an inter-CHU multicenter study as well as the creation and provision of a database (cohort) for artificial intelligence procedures.

ELIGIBILITY:
Inclusion Criteria:

* Bimaxillary edentulous patients
* Former bimaxillary CRP wearers (transitional or usage)
* Acceptance of the confiscation of the old prosthesis when the new prosthesis is placed in the mouth and during the 4 months the new prosthesis is worn.
* Signed informed consent

Exclusion Criteria:

* Dependent patients (under guardianship or patients in EHPAD)
* Heavy pathologies
* Salivary pathologies (Gougerot-Sjögren syndrome) or asialia related to a medication.
* Patients with a pacemaker
* Skeletal class III with an anteroposterior shift of more than 1 cm
* Patients under court protection

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-25 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
masticatory muscle activity at 1 month of wearing prostheses | 1month
  Measurement of muscle activity = measurements will be made for all muscles at rest with and without prostheses.
masticatory muscle balance at 1 month of wearing prostheses | 1month
  Muscle balance analysis = comparison of right and left muscle activity.

SECONDARY OUTCOMES:
number of sessions required to obtain a finalized prosthesis | 1 month
  The number of sessions required to obtain a finalized prosthesis recorded for each patient is listed.
quality of life of the patients at 1 month of wearing the prosthesis | 1 month
  The quality of life of the patients is assessed using a specific oral health measurement questionnaire (GOHAI). The GOHAI includes 12 items with 3 sub-dimensions (functional, psycho-social and pain/discomfort).
  For each assessment (inclusion visit, 1-month post completion visit and 4-month post completion visit), the 3 sub-dimensions will be analyzed.
  The patient must answer the 12 questions with "Never", "Rarely", "Sometimes", "Often" or "Always" (only one answer possible). Each answer is scored from 5 to 1 in this order, except for questions 3, 5 and 7 where the values are reversed. The associated total score varies from 12 to 60. The higher the score, the better the oral quality of life. The score obtained is classified into three categories:
  12< <50: poor oral quality of life 51< <56: average oral quality of life 57< <60: good oral quality of life
quality of life of the patients at 4 months of wearing the prosthesis | 4 months
  The quality of life of the patients is assessed using a specific oral health measurement questionnaire (GOHAI). The GOHAI includes 12 items with 3 sub-dimensions (functional, psycho-social and pain/discomfort).
  For each assessment (inclusion visit, 1-month post completion visit and 4-month post completion visit), the 3 sub-dimensions will be analyzed.
  The patient must answer the 12 questions with "Never", "Rarely", "Sometimes", "Often" or "Always" (only one answer possible). Each answer is scored from 5 to 1 in this order, except for questions 3, 5 and 7 where the values are reversed. The associated total score varies from 12 to 60. The higher the score, the better the oral quality of life. The score obtained is classified into three categories:
  12< <50: poor oral quality of life 51< <56: average oral quality of life 57< <60: good oral quality of life
masticatory muscle activity at the insertion of prostheses in mouth | at the insertion of prostheses in mouth
  Measurement of muscle activity = measurements will be made for all muscles at rest with and without prostheses.
masticatory muscle activity at 4 months of wearing prostheses | 4 months
  Measurement of muscle activity = measurements will be made for all muscles at rest with and without prostheses.
masticatory muscle balance at the insertion of prostheses in mouth | at the insertion of prostheses in mouth
  Muscle balance analysis = comparison of right and left muscle activity.
masticatory muscle balance at 4 months of wearing prostheses | 4 months
  Muscle balance analysis = comparison of right and left muscle activity.
Analysis of the chronology of muscle contraction on the right and left | 1 month
  Analysis of the chronology of muscle contraction on the right and left = muscle contraction symmetry

CONTACTS AND LOCATIONS:
Overall Officials: Delphine Carayon, MCU-PH, Principal Investigator — University Hospital, Montpellier
Locations (1):
- CHU de Montpellier, Montpellier, France